CLINICAL TRIAL: NCT00351195
Title: A Phase II Study of Etoposide, Oxaliplatin and Capecitabine in Patients With Advanced HCC
Brief Title: Etoposide, Oxaliplatin and Capecitabine in Advanced Hepatocellular Carcinoma (HCC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not meet the criteria for continuation to second stage
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Morten Ladekarl, MD, DMSc., Dept. of Oncology, Århus Sygehus, Århus (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: etoxel-01-2005
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Etoposide; Oxaliplatin; Capecitabine
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Etoposide; Oxaliplatin; Capecitabine

INTERVENTIONS:
Drug: Etoposide
Drug: Oxaliplatin
Drug: Capecitabine

SUMMARY:
Various cytotoxic agents have been evaluated in advanced hepatocellular carcinoma, but response rates have been low with significant toxicity, most often due to parenchymal liver disease. The three agents etoposide, oxaliplatin and capecitabine each has sparse efficacy as single agents, but the combination may act synergistically with an acceptable toxicity profile.

DETAILED DESCRIPTION:
Design:

Open phase II study.

Purpose:

Response rate for the combination of etoposide, oxaliplatin and capecitabine given every 3 weeks on an outpatient basis.

Secondary endpoint are safety, time to progression and survival

Treatment:

Etoposide are administered intravenously 100 mg/m2 on day 1 and orally 200 mg/m2 on days 2 and 3.

Capecitabine (Xeloda) are administered 1000 mg/m2 twice daily with 12 hours interval for two weeks and one week off

Oxaliplatin are administered intravenously 100 mg/m2 on day 1 in each cycle as a 2 hours infusion.

One cycle is 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified intra- or extrahepatic inoperable hepatocellular carcinoma or hyperdense liver lesion at computed tomography and concurrent elevated alpha-feto-protein > 400 ng/ml
* PS 0-2
* Age 18-75
* Life expectancy > 12 weeks
* Normal bone marrow function (neutrophiles > 1,5 x 109/l and platelets > 100 x 109/l)
* Bilirubin < 2 x UNL
* Transaminases < 3 x UNL
* Normal renal function, Cr-EDTA clearance > 50 ml/min
* No chemotherapy, radiotherapy or immunotherapy 4 weeks prior to inclusion
* No uncontrolled, severe concurrent medical disease
* Fertile women must have a negative pregnancy test
* Fertile women must use adequate contraceptives during and 3 months after trial exposure
* Signed informed consent

Exclusion Criteria:

* Chemotherapy, radiotherapy or immunotherapy 4 weeks prior to inclusion
* Experimental therapy < 8 weeks prior to inclusion
* Known DPD-deficiency
* Known neuropathy
* Uncontrolled, severe concurrent medical disease
* Prior malignancy during the last 5 years, except for non-melanoma skin cancer and carcinoma in situ cervix uteri.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2006-02; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Response

SECONDARY OUTCOMES:
Time to progression
Safety
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Lassen, MD., PH.D., Principal Investigator — Rigshospitalet, Dept. of Oncology
Locations (1):
- Århus Sygehus, Dept. of Oncology, Aarhus, Denmark